CLINICAL TRIAL: NCT02153684
Title: Canadian Cohort on the Origin and Progression of Airway Disease: Physiology Platform
Status: Completed | Type: Observational
Sponsor: Dr. Denis O'Donnell (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ottawa Hospital Research Institute (Other); University of British Columbia (Other); McGill University (Other)
Responsible Party: Sponsor-Investigator, Dr. Denis O'Donnell, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Other Study IDs: DMED-1674-14
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Smoking; COPD
Keywords: smoking; small airway dysfunction; mild COPD; dyspnea; exercise; clinical outcomes
MeSH Terms: conditions — Smoking; Pulmonary Disease, Chronic Obstructive; Dyspnea; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Mild COPD, symptomatic: Smokers fitting GOLD 1B criteria for COPD
- Mild COPD, asymptomatic: Smokers fitting GOLD 1A criteria for COPD
- Symptomatic smokers, at risk for COPD: Smokers who do not meet spirometric criteria for COPD
- Healthy, non-smoking controls: Non-smokers, matched to smoking groups for age (>40 yrs of age) and gender

SUMMARY:
The Canadian Respiratory Research Network (CRRN) has recently been established to study the origins and evolution of airways disease in the population. The CRRN is funded by the Institute of Cardio-respiratory Health (ICRH), an institute of the CIHR. The Physiology platform will support the other CRRN platforms (biology, imaging, population health, knowledge transfer) by providing a comprehensive characterization of the nature and extent of physiological impairment of respiratory function in smokers at risk for airways disease and in those with early or mild airway obstruction. The planned studies of the physiology group (core sites located at Queen's University, University of British Columbia and McGill University) will initially focus on smoking-related lung injury in those at risk for COPD and in those meeting spirometric criteria for mild airway obstruction, with or without respiratory symptoms. The primary aim of this initial study is to identify and validate sensitive test(s) of peripheral airway dysfunction that may qualify as physiological biomarkers for use in future CRRN studies.

ELIGIBILITY:
INCLUSION CRITERIA:

Stable patients with GOLD grade 1 mild COPD will be included in the study if they have: a post-bronchodilator FEV1≥80 %predicted and an FEV1/FVC ratio <0.7 and <LLN; ≥40 years of age; and a cigarette smoking history ≥10 pack-years or ≥10 years of exposure to other inhaled substances (i.e., second hand smoke and/or biomass). Symptomatic (category B) subjects will have a Baseline Dyspnea Index (BDI) total score ≤9, a modified Medical Research Council (MRC) dyspnea score ≥2, or a COPD Assessment Test (CAT) score ≥10. Asymptomatic (category A) subjects will have a BDI>9, modified MRC<2 or CAT<10, no history of seeking medical care for respiratory symptoms, and no history of using respiratory medications. Symptomatic current or ex-smokers (>10 pack-year history) who do not meet criteria for COPD (e.g., post-bronchodilator FEV1<80%predicted and FEV1/FVC<0.7, with both measurements also <LLN) and who are on no respiratory medication will be included. Symptomatic will be defined as: BDI≤9, modified MRC≥2 or CAT>10. Healthy, age- and sex-matched, non-smoking (<2 pack-year history) participants with normal spirometry will be used for comparison purposes.

EXCLUSION CRITERIA:

* presence of clinically significant comorbidities that could contribute to dyspnea or exercise limitation (i.e., unstable heart disease, a pulmonary disease other than COPD, uncontrolled diabetes, neuromuscular or orthopedic impairment);
* history/clinical evidence of asthma;
* contraindications to exercise testing;
* <40 years of age;
* body mass index <18.5 or >=35 kg/m2.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will include 30 participants from each of the following four subgroups: GOLD grade 1A COPD, GOLD grade 1B COPD, symptomatic smokers who do not meet spirometric criteria for COPD, and age- and sex-matched healthy non-smoking controls. Subjects will be recruited from the Canadian Chronic Obstructive Lung Disease (CanCOLD) study cohort and, once that source has been exhausted, from each site's database of previous or potential research study participants. The CanCOLD Study cohort was recruited from the COLD Study sample, which was a random sample of adults ≥40 years of age who had pre- and post-bronchodilator spirometry performed in order to estimate the prevalence of COPD in Canada.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Small airway function | 1 day (Time of visit)
  There is no single measurement of small airway function since this study is evaluating which measurements, among a list of conventional and experimental physiological parameters, best characterize the nature and extent of impairment of respiratory function in the smoking study groups and which of these parameters best predict clinical outcome (i.e., dyspnea, exercise capacity, ventilatory capacity, health status). Assessments will include: spirometry, closing volume, impulse oscillometry, frequency dependence of dynamic lung compliance, plethysmographic lung volumes and metronome-paced dynamic hyperinflation.

SECONDARY OUTCOMES:
Cardiopulmonary exercise test | 1 day (Time of visit)
  Includes measurements of exertional dyspnea (intensity and quality), peak exercise capacity (peak oxygen uptake [VO2]) and ventilatory responses (ventilation, pulmonary gas exchange, breathing pattern, operating lung volumes and tidal flow-volume loops) during symptom-limited incremental cardiopulmonary cycle exercise testing.
Clinical outcome | 1 day (Time of visit)
  Includes questionnaires regarding chronic activity-related dyspnea, respiratory symptoms, health status and physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, FRCPC, Principal Investigator — Queen's University and Kingston General Hospital
Locations (3):
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - Queen's University and Kingston General Hospital, Kingston, Ontario
  - McGill University, Montreal, Quebec